CLINICAL TRIAL: NCT00604058
Title: Immunogenicity and Safety of Fractional Doses of Sanofi Pasteur's Inactivated Poliomyelitis Vaccine Administered Intradermally vs Full Doses of Inactivated Poliomyelitis Vaccine Administered Intramuscularly in Healthy Philippines Infants
Brief Title: Immunogenicity and Safety of Fractional Doses of IPV Intradermally vs Full Doses Intramuscularly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV25
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Poliomyelitis
Keywords: Poliomyelitis; intradermal
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated; Rabies Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Inactivated Poliomyelitis vaccine (IMOVAX)
- Group B (Active Comparator)
  Interventions: Biological: Inactivated Poliomyelitis vaccine (IMOVAX)

INTERVENTIONS:
Biological: Inactivated Poliomyelitis vaccine (IMOVAX) — Fractional dose (1/5th) 0.1 mL, intradermally
  Other Names: IMOVAX Polio (IPV) vaccine
  Arms: Group A
Biological: Inactivated Poliomyelitis vaccine (IMOVAX) — A full dose, 0.5 mL, intramuscular
  Other Names: IMOVAX Polio (IPV) vaccine
  Arms: Group B

SUMMARY:
The present study intends to investigate the use of fractional doses of sanofi pasteur's IMOVAX Polio injected intradermally. The primary objective will be to demonstrate the non-inferiority of fractional doses of IMOVAX Polio administered intradermally versus full doses of IMOVAX Polio administered intramuscularly, in terms of seroprotection rates (polio types 1, 2 and 3) one month after the three-dose primary vaccination administered at 6-10-14 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria to be checked at the screening visit (SC):
* Aged 0 to 7 days on the day of screening
* Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥2.5 kg
* Informed consent form signed by the parent(s) or other legally acceptable representative
* Subjects and parent/guardian able to attend all scheduled visits and comply with all trial procedures
* Inclusion Criteria to be checked at the randomization visit (V01):
* Aged 42 to 50 days on the day of inclusion
* Subjects and parent/guardian able to attend all scheduled visits and comply with all trial procedures

Exclusion Criteria:

* Exclusion Criteria to be checked at the screening visit (SC):
* Planned participation in another clinical trial during the present trial period
* Illness that could interfere with trial conduct or completion, in the opinion of the investigator
* Receipt of blood or blood-derived products since birth that might interfere with the assessment of immune response
* History of seizures
* Known personal or maternal Human Immunodeficiency Virus (HIV), Hepatitis B antigen or Hepatitis C seropositivity
* Thrombocytopenia or bleeding disorder contraindicating IM injection
* Exclusion Criteria to be checked at the randomization visit (V01):
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Receipt of blood or blood-derived products since birth that might interfere with the assessment of immune response
* Receipt or planned receipt of any vaccine in the 4 weeks preceding or following any trial vaccination (except BCG, DTP-Hib or Hepatitis B vaccines, which can not be given within 10 days before or after any study vaccination)
* History of seizures
* Known personal or maternal Human Immunodeficiency Virus (HIV), Hepatitis B antigen or Hepatitis C seropositivity
* History of poliomyelitis infection (confirmed either clinically, serologically or microbiologically)
* Previous vaccination against the poliomyelitis disease with either the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular (IM) injection
* Febrile illness (temperature ≥38°C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment

Ages: 42 Days to 50 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The non-inferiority of fractional doses of IMOVAX Polio administered intradermally versus full doses of IMOVAX Polio administered intramuscularly, in terms of seroprotection rates (polio types 1 2 and 3) one month after the three-dose primary vaccination | 1 Month Post-vaccination

SECONDARY OUTCOMES:
Immunogenicity: To assess and describe in each group the immunogenicity of the study vaccines one month after the three-dose primary vaccination Safety: To describe in each group the safety after each dose of the study vaccines | 1 Month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- Quezon City, Manila, Philippines

REFERENCES:
- [Derived] Cadorna-Carlos J, Vidor E, Bonnet MC. Randomized controlled study of fractional doses of inactivated poliovirus vaccine administered intradermally with a needle in the Philippines. Int J Infect Dis. 2012 Feb;16(2):e110-6. doi: 10.1016/j.ijid.2011.10.002. Epub 2011 Dec 5. PMID 22153001
- See also: Related Info — http://www.sanofipasteur.com